CLINICAL TRIAL: NCT06183996
Title: Patterns Of Floppy Infants Attending Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christina Sameh Youssef Ghaly, Assistant Lecturer, Assiut University
Other Study IDs: CS
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Floppy Infant
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The Floppy Infant includes a variety of signs and symptoms: hypotonia, weakness and ligamentous laxity and increased range of joint mobility. Based on clinical criteria hypotonia can be classified in two major groups: central and peripheral hypotonia .The primary objective of the diagnosis is to enable an early identification of the problem to start an effective supportive therapy. Also allows formulating a more accurate prognosis. Last, the identification of forms of neonatal hypotonia with familial transmission is crucial for genetic counseling for future pregnancies.etiology in hypotonic infants is necessary for prognosis prediction and treatment. History taking and physical examination should be supported by the laboratory tests and neuroimaging methods. However, diversity may require a genetic diagnosis.

DETAILED DESCRIPTION:
The Floppy Infant includes a variety of signs and symptoms: decrease in muscle tone (hypotonia), in muscle power (weakness) and ligamentous laxity and increased range of joint mobility. Based on clinical criteria hypotonia can be classified in two major groups: central hypotonia and peripheral hypotonia .

Hypotonia is defined as poor muscle tone in the muscles of the trunk, limbs and face. This means that the muscles provide little resistance when someone else is passively moving them. Hypotonia can be categorized as axial or truncal ,predominantly affecting the neck and spinal muscles; appendicular, affecting predominantly the extremities; or global, affecting the entire body. It is identified early in life when the newborn is unable to obtain a normal posture during movements or at rest.

Regardless of whether the underlying cause of hypotonia is peripheral or central in origin, the presentation of floppy infant syndrome focuses on observing for the presence or absence of specific signs such as 'frog-leg' posture, significant head lag on traction or pull-to-sit maneuver, or the feeling of 'slipping through the hands' when the infant is held under the arms.

The primary objective of the diagnosis is to enable, where possible, an early identification of the problem to start an effective supportive therapy. A precise etiological diagnosis also allows formulating a more accurate prognosis. Last but not least, the identification of forms of neonatal hypotonia with familial transmission is crucial for the formulation of a genetic counseling for future pregnancies.

Inspite of the advances in laboratory diagnosis and imaging, multidisciplinary evaluation by different specialties including genetics, metabolics , pediatric neurology and pediatric neuroradiology is mandatory .

sometimes, the etiology cannot be found. Although it is difficult to define the underlying etiology in hypotonic infants, it is necessary to know the etiology for prognosis prediction and treatment. History taking and physical examination should be supported by the laboratory tests and neuroimaging methods. However, diversity may require a genetic diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Infants presented by generalized hypotonia and hyporeflexia

Exclusion Criteria:

* Infants with global developmental delay & Central causes of hypotonia

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants presented by generalized hypotonia and hyporeflexia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Patterns Of Floppy Infants Attending Assiut University Children's Hospital | 2 years
  Evaluate the percentage of floppy infants with peripheral causes in relation to the whole cases of floppy infants attending Assiut university children hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahrous El Tallawy, Professor, Study Chair — Assiut University; Eman Fathalla Gad, Assistant Professor, Study Director — Assiut University; Mohamed Abo bakr Mohamed, Lecturer, Study Director — Assiut University